CLINICAL TRIAL: NCT05313503
Title: KETOMIGRAINE: "Ketogenic Diet in Patients With Drug-resistant Chronic Migraine, "Non-responder" to Treatment With Monoclonal Antibody Targetting CGRP Pathway: a Pilot Study, Open Label"
Brief Title: KETOMIGRAINE: Ketogenic Diet in Drug-resistant Chronic Migraineurs
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KETOMIGRAINE2021
Record Dates: First submitted 2022-03-11; First posted 2022-04-06 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-03

CONDITIONS: Chronic Migraine, Headache
Keywords: Ketogenic Diet; reistant migraine; CGRP; headache; pain
MeSH Terms: conditions — Headache; Pain | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: interventional, monocentric, open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ketogenic Diet (Experimental): Ketogenic diet
  Interventions: Other: ketogenic diet

INTERVENTIONS:
Other: ketogenic diet — We propose a type of KD named MAD (Modified Atkins Diet) characterized by the following percentages of macronutrients: 65% fats, 27% proteins and 8% carbohydrates.

SUMMARY:
Our protocol, named "KETOMIGRAINE", is based on the prescription of a Ketogenic Diet (KD) to twenty subjects with diagnosis of Chronic Migraine (CM), resistant to oral preventive treatments and non-responders to monoclonal antibodies targeting the CGRP pathway. The trial starts with one month of baseline during which are verified inclusion/exclusion criteria. After that, participants will assume KD for three months, a transitional diet (TD) for other three months. Follows a period of three months of free diet (FD). Neurological and dietician visits are scheduled during the course of the trial.

DETAILED DESCRIPTION:
The duration of the trial for individual participants is approximately 10 months, divided as follows: 1 month of baseline + 3 months of KD + 3 months of TD+ 3 months of follow-up.

The protocol includes 6 neurological evaluations (T0-T5); 11 dietary evaluations, some of which can be remote visits, and will be defined below with the acronym "V" (V1-V11).

The planned activities are listed below:

* T0 screening: neurological and general physical examination, extended anamnestic evaluation, evaluation of the inclusion / exclusion criteria. Signature of the informed consent for participation in the research study, assignment of an identification code (increasing number starting from 01); headache diary delivery for prospective baseline data collection.
* T1 baseline (30 days +/- 3 after T0): assessment of compliance in filling in the headache diary and confirming the diagnosis of chronic migraine; execution of electrocardiogram, pregnancy test (if female patient with childbearing potential) and blood tests (renal, hepatic, lipidic, endocrinological profile); first dietary visit (V1 - anthropometric measurements-BMI, interview on eating habits), nutritional instrumental evaluations (calorimetry and body composition).
* T2 Day 1 (Enrollment -7 days +/- 3 after T1): verification of inclusion and exclusion criteria with the results of blood tests; blood sample for collection of PACAP, CGRP and metabolites of kynurenines; compilation of the disability and impact questionnaires - MIDAS and HIT-6; compilation of Migraine Specific Quality of Life Questionnaire (MSQ); dietary assessment (V2): prescription of the KD that the patient will follow for the next 3 months. Subjects overweight will follow a KD with a low-calorie content (low-calorie ketogenic diet); patients with a lower BMI will follow a normo-caloric diet: those represent the two subgroups of the study. Both subtypes of diet (normo and low-calorie) will induce at the same way ketosis; the only difference between the two subgroups is the fact that one will be associated with weight loss and the other not. During the three months of KD, dietician evaluations will be carried out every two weeks, alternating those remotely with those onsite (V3-V7). The dietary visits at the end of the 1st, 2nd and 3rd month of KD will be carried out onsite and the ketone dosage will be carried out using blood sticks.
* T3 (3 months from T2 - end of KD and start of transitional diet - TD): evaluation of the headache diary and compilation of the disability and impact scales - MIDAS and HIT-6); repetition of blood tests in order to check dietary tolerance; blood sample for CGRP, PACAP, metabolites of kynurenines (II point); repetition of instrumental measurements (calorimetry and body composition); dietary visit (V8) for the last check of ketonemia and prescription of TD. This type of diet is not ketogenic and is characterized by the gradual introduction of carbohydrates starting from breakfast, it will last for 3 months. Onsite dietary visits (V9-V10) follow on a monthly basis
* T4 (3 months after T3 - end of TD and start of free diet - FD): neurological and dietary visit (V 11) at the end of 3 months of TD. The patient will start a free diet, during which he/she can eat what is preferred.
* T5 (3 months after T4 - end of study): The last visit is a follow-up, 9 months after T2, its purpose is to evaluate the trend of headache parameters, BMI and biochemical markers studied (III point). During this visit will be filled the following questionnaires: disability and impact questionnaires - MIDAS and HIT-6, Migraine Specific Quality of Life Questionnaire (MSQ), Patient's Global Impression of Change (PGIC).

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-65 years old
* Chronic migraine, diagnosed according to ICHD-3 criteria.
* Patients with resistant form of migraine defined as: persistence of 8 days of headache per month; therapeutic failure (after therapeutic treatment of adequate dose and duration) or contraindication of 3 classes of drugs with validated evidence of efficacy in the prevention of migraine.
* Non-responder (absence of reduction of MIDAS score of at least 50% after at least 3 months of treatment) to at least one anti-CGRP monoclonal antibody
* Absence of prophylactic therapies for migraine or prophylaxis therapy with a single drug taken at a stable dose for at least two months
* BMI > 16.5 kg/m2 and < 35 kg/m2
* Hypothesized compliance in filling the headache diary and following the prescribed diet

Exclusion Criteria:

* Kidney failure
* Liver failure
* Heart failure
* Recent heart attack
* Pancreatitis
* Alcoholism
* Severe osteoporosis
* Other neurological disorders, including other forms of primary headache, except sporadic episodic tension-type headache
* Diabetes Mellitus
* Severe lipid metabolism disorders
* Women of childbearing age without active contraception
* Pregnancy or breastfeeding
* Psychiatric disorders that the clinician thinks may interfere with patient compliance / eating disorders
* Other anomalies considered significant in preliminary examinations (blood tests and EKG)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Change of mean monthly migraine days | During the 3 months of Ketogenic diet period
  The primary endpoint is the change of mean monthly migraine days during the treatment phase compared to the baseline period. The number of migraine days will be established by the analysis of the headache diary that the patients are required to fill in for the duration of the study

SECONDARY OUTCOMES:
Change of number of headache day per month | Through study completion, an average of 10 months
  Evaluation of the change of headache day per month during the study. The number of headache days will be established by the analysis of the headache diary that the patients are required to fill in for the duration of the study
Change of doses of symptomatic drug intake per month | Through study completion, an average of 10 months
  Evaluation of the change of doses of symptomatic drug intake per month. The number of doses of symptomatic drug intake days will be established by the analysis of the headache diary that the patients are required to fill in for the duration of the study
Change of number of days of moderate to severe headache | Through study completion, an average of 10 months
  Evaluation of the change of days of moderate to severe headache during the study. The number of moderate to severe headache days will be established by the analysis of the headache diary that the patients are required to fill in for the duration of the study
Change of days of symptomatic drug intake per month | Through study completion, an average of 10 months
  Evaluation of the change of days of symptomatic drug intake per month. The number of days of symptomatic drug intake days will be established by the analysis of the headache diary that the patients are required to fill in for the duration of the study
Change of average pain intensity | Through study completion, an average of 10 months
  Evaluation of the change of average pain intensity during the study. The average pain intensity will be established by the analysis of the headache diary that the patients are required to fill in for the duration of the study
change in disability of headache | Through study completion, an average of 10 months
  Evaluation of the change in disability of headache by measuring the variation in points of the questionnaire filled out by the patient named MIDAS (Migraine Disability Assessment). It has 5 items and evaluates the disability caused by headache. A higher score means more disability caused by headache.
change in impact of headache | Through study completion, an average of 10 months
  Evaluation of the change in impact of headache by measuring the variation in points of the questionnaire filled out by the patient named HIT-6 (Headache Impact Test-6). It has 6 item and evaluates the impact of headache on routinary activities. A higher score means more impact caused by headache.
change in total pain burden | Through study completion, an average of 10 months
  The purpose is to evaluate the change in total pain burden (number of hours of headache * pain intensity on a scale from 1 to 3) over three months of the KD. These data are established by the analysis of the headache diary hat the patient fills out during all the protocol phases.
change in quality of life | Through study completion, an average of 10 months
  The change in quality of life is evalueted through the administration of questionnare named: "Migraine Specific Quality of Life Questionnaire" (MSQ) that has 14 items. High score means higher influence of migraine in daily activities.
Patient's Global Impression of Change | Through study completion, an average of 10 months
  The patients impression of change is evaluated with the administration of a questionnaire: "Patient's Global Impression of Change (PGIC)" that has 1 item with 7 answer options, the seventh option is the best impression of change.
Evaluation of persistence of KD benefits | Through study completion, an average of 10 months
  The persistence of KD benefits after a period of follow-up is measured by processing the difference in monthly migraine days at the end of follow-up compared to migraine days during KD.
Mechanism of action of KD | During the 3 months of Ketogenic diet period
  In-depth comprehension of the mechanism of action of KD by evaluating the variation of the plasma levels of neuropeptides involved in the pathophysiology of migraine (Calcitonin Gene Related Peptide CGRP and Peptide Activating Adenylate Cyclase of the Pituitary - PACAP) and of some metabolites of kynurenines (kynurenic and quinolinic acid). These data are obtained by blood samplings.

OTHER OUTCOMES:
Effect of KD in the subgroups identified by the type of diet (normal-calorie and low-calorie diet) | Through study completion, an average of 10 months
  The exploratory outcome is to describe the effect of KD in the subgroups identified by the type of diet (normal-calorie and low-calorie diet) in terms of difference of headache days' reduction / per month; the data will be obtained with the analysis of the headache diary filled by the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, Prof, Study Director — IRCCS Mondino Foundation, Pavia
Locations (1):
- Headache Science Center, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] de Almeida Rabello Oliveira M, da Rocha Ataide T, de Oliveira SL, de Melo Lucena AL, de Lira CE, Soares AA, de Almeida CB, Ximenes-da-Silva A. Effects of short-term and long-term treatment with medium- and long-chain triglycerides ketogenic diet on cortical spreading depression in young rats. Neurosci Lett. 2008 Mar 21;434(1):66-70. doi: 10.1016/j.neulet.2008.01.032. Epub 2008 Jan 19. PMID 18281154
- [Result] Di Lorenzo C, Coppola G, Sirianni G, Di Lorenzo G, Bracaglia M, Di Lenola D, Siracusano A, Rossi P, Pierelli F. Migraine improvement during short lasting ketogenesis: a proof-of-concept study. Eur J Neurol. 2015 Jan;22(1):170-7. doi: 10.1111/ene.12550. Epub 2014 Aug 25. PMID 25156013
- [Result] Bongiovanni D, Benedetto C, Corvisieri S, Del Favero C, Orlandi F, Allais G, Sinigaglia S, Fadda M. Effectiveness of ketogenic diet in treatment of patients with refractory chronic migraine. Neurol Sci. 2021 Sep;42(9):3865-3870. doi: 10.1007/s10072-021-05078-5. Epub 2021 Feb 1. PMID 33527209